CLINICAL TRIAL: NCT04005001
Title: Using Clinical Treatment Data in a Machine Learning Approach for Sepsis Detection
Brief Title: Machine Learning Sepsis Alert Notification Using Clinical Data
Acronym: HindSight P2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dascena (Industry)
Collaborators: Cape Regional Medical Center (Unknown); Cooper University Medical Center (Unknown); Baystate Health (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-569185; 2R44AA030000-02 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Sepsis; Machine learning algorithm; Clinical decision support
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — peb protein, Drosophila; Compact Disks; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental arm will involve patients monitored by HindSight.
  Interventions: Other: HindSight
- Control (Active Comparator): The control arm will involve patients monitored by InSight.
  Interventions: Other: InSight

INTERVENTIONS:
Other: HindSight — HindSight will examine the dynamic trends of clinical measurements taken from a patient's EHR and analyzes correlations between vital signs to alert for the onset of sepsis.This machine learning based tool is optimized by encoder and utilizes periodic retraining to improve its performance over time.
  Other Names: HindSight-Clinical decision support (CDS) system for sepsis alert notification
  Arms: Experimental
Other: InSight — Compared to the ability of the InSight software's recognition of sepsis onset to HindSight's performance. The study determines if the HindSight software has equivalent or better performance than the InSight software.
  Arms: Control

SUMMARY:
Machine learning is a powerful method to create clinical decision support (CDS) tools, when training labels reflect the desired alert behavior. In our Phase I work for this project, we developed HindSight, an encoding software that was designed to examine discharged patients' electronic health records (EHRs), identify clinicians' sepsis treatment decisions and patient outcomes, and pass those labeled outcomes and treatment decisions to an online algorithm for retraining of our machine-learning-based CDS tool for real-time sepsis alert notification, InSight. HindSight improved the performance of InSight sepsis alerts in retrospective work. In this study, we propose to assess the clinical utility of HindSight by conducting a multicenter prospective randomized controlled trial (RCT) for more accurate sepsis alerts.

DETAILED DESCRIPTION:
We will evaluate the performance of HindSight in a randomized controlled trial (RCT). HindSight is a novel encoding software designed to optimize alerts for sepsis alert notification. HindSight identifies clinicians' sepsis-related decisions in the electronic health records of former patients and passes those events to InSight, thus supplying InSight with labeled examples of true positive sepsis cases for retraining. In our retrospective work, we have shown that HindSight enables InSight to adapt to site-specific deviations of real-world clinical deployment by successfully reducing false and irrelevant alarms, without human supervision. The goal of this project is to demonstrate that the retrospective success of HindSight can be successfully translated to live clinical environments. In our Phase I work, HindSight achieved an area under the receiver-operating characteristic (AUROC) of 0.899, 0.831 and 0.877 for clinician sepsis evaluation, treatment, and onset, respectively. By using an online learning algorithm to incorporate HindSight-labeled data into the InSight predictor, we showed that the online-trained InSight can adapt to the HindSight-labeled data and outperform both baseline and periodically re-trained versions of InSight (p < 0.05). In Aim 1, we will prospectively validate HindSight's performance on real-time patient data streams in three diverse hospitals non-interventionally. In Aim 2, we will evaluate the effect of the tool in a prospective, interventional RCT. HindSight will first be evaluated by live deployment at four academic and community hospitals, during which time it will not provide alerts of future sepsis onset. Following any necessary algorithm optimization arising from live hospital validation, we will perform an RCT to evaluate reductions in false alerts from InSight trained on HindSight sepsis labels (experimental arm), compared to InSight trained on gold standard Sepsis-3 labels (control arm).

ELIGIBILITY:
Inclusion Criteria:

* During the study period, all patients over the age of 18 presenting to the emergency department or admitted to an inpatient unit at the participating facilities will automatically be enrolled in the study, until the enrollment target for the study is met

Exclusion Criteria:

* Patients under the age of 18
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37986 (Estimated)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of reduction in false alerts | Through study completion, human subjects involvement will occur for an average of eight months
  The primary outcome measure of interest will be false alert reduction. Successful completion of Aim 1 will be demonstrated by a positive predictive value (PPV) in a live clinical setting for which the lower bound of the 95% confidence interval meets or exceeds the benchmark from prior retrospective studies. Meeting the retrospective PPV benchmark indicates that prospective CDS quality reflects retrospective CDS quality, and is sufficiently high to reduce alarm fatigue and improve clinical utility. Success of Aim 2 is contingent upon achieving a 15% relative reduction in false alerts when comparing between the two treatment arms (p < 0.05; Fisher's Exact Test).

CONTACTS AND LOCATIONS:
Overall Officials: Jana Hoffman, PhD, Principal Investigator — Dascena
Locations (3):
- United States (3):
  - Baystate Health, Springfield, Massachusetts
  - Cooper University Health Care, Camden, New Jersey
  - Cape Regional Medical Center, Cape May, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desautels T, Calvert J, Hoffman J, Mao Q, Jay M, Fletcher G, Barton C, Chettipally U, Kerem Y, Das R. Using Transfer Learning for Improved Mortality Prediction in a Data-Scarce Hospital Setting. Biomed Inform Insights. 2017 Jun 12;9:1178222617712994. doi: 10.1177/1178222617712994. eCollection 2017. PMID 28638239
- [Background] Calvert J, Mao Q, Rogers AJ, Barton C, Jay M, Desautels T, Mohamadlou H, Jan J, Das R. A computational approach to mortality prediction of alcohol use disorder inpatients. Comput Biol Med. 2016 Aug 1;75:74-9. doi: 10.1016/j.compbiomed.2016.05.015. Epub 2016 May 24. PMID 27253619
- [Background] Calvert JS, Price DA, Barton CW, Chettipally UK, Das R. Discharge recommendation based on a novel technique of homeostatic analysis. J Am Med Inform Assoc. 2017 Jan;24(1):24-29. doi: 10.1093/jamia/ocw014. Epub 2016 Mar 28. PMID 27026611
- [Background] Calvert J, Mao Q, Hoffman JL, Jay M, Desautels T, Mohamadlou H, Chettipally U, Das R. Using electronic health record collected clinical variables to predict medical intensive care unit mortality. Ann Med Surg (Lond). 2016 Sep 6;11:52-57. doi: 10.1016/j.amsu.2016.09.002. eCollection 2016 Nov. PMID 27699003
- [Background] Shimabukuro DW, Barton CW, Feldman MD, Mataraso SJ, Das R. Effect of a machine learning-based severe sepsis prediction algorithm on patient survival and hospital length of stay: a randomised clinical trial. BMJ Open Respir Res. 2017 Nov 9;4(1):e000234. doi: 10.1136/bmjresp-2017-000234. eCollection 2017. PMID 29435343